CLINICAL TRIAL: NCT00065195
Title: Efficacy of Massage at the End of Life
Brief Title: REST: Reducing End-of-Life Symptoms With Touch
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT001006-01A2 (NIH)
Record Dates: First submitted 2003-07-18; First posted 2003-07-21 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Neoplasms; Pain
Keywords: Massage; Palliative Care; Hospices; Cancer
MeSH Terms: conditions — Neoplasms; Pain

INTERVENTIONS:
Procedure: Moving touch therapy
Procedure: Nonmoving touch therapy

SUMMARY:
The purpose of this study is to determine whether massage therapy is effective in reducing pain and distress and improving quality of life among cancer patients at life's end.

DETAILED DESCRIPTION:
Relieving physical and emotional symptoms is a key component of end-of-life care. Despite care, terminally ill patients are still significantly burdened by unrelieved symptoms. Therapies that have potential to alleviate these symptoms deserve thorough investigation.

This study will last 3 weeks. Participants in this study will be randomly assigned to receive six sessions of either moving or nonmoving touch therapy, in addition to usual hospice care, for 2 weeks. Moving touch therapy consists of massage therapy in which a trained therapist continually touches a person's body. The nonmoving touch therapy will be conducted by volunteers who have no previous experience in massage. Participants in this group will have a volunteer rub specific body parts for 3-minute intervals. Because current evidence suggests that thoughts of healing may influence the effectiveness of touch therapy, volunteers in the nonmoving therapy group will distract their minds to avoid thinking of healing processes. In both groups, the person administering the touch therapy will note all interruptions during a session, including talk, music, and television. Interviews about medication use, pain, and quality of life will be used to assess participants; these interviews will be conducted at study start, immediately before and after each therapy session, and at Weeks 1, 2, and 3.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer, with at least moderate pain 1 week prior to study entry
* Life expectancy of at least 3 weeks
* Able to speak English

Exclusion Criteria:

* Massage therapy within 1 month prior to study entry
* Current use of anticoagulants
* Platelet count less than 10,000
* Unstable spine that would interfere with touch therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440
Dates: Start 2003-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Decreased pain

SECONDARY OUTCOMES:
Less total analgesic medication use.
Improved quality of life
Decreased physical symptom distress
Decreased emotional symptom distress

CONTACTS AND LOCATIONS:
Overall Officials: Jean S. Kutner, MD, Principal Investigator — University of Colorado, Denver; Marlaine Smith, RN, PhD, Principal Investigator — University of Colorado, Denver
Locations (9):
- United States (9):
  - San Diego Hospice, San Diego, California
  - Pike's Peak Hospice and Palliative Care, Colorado Springs, Colorado
  - Pathways at Hospice of Metro Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Hospice of St. John, Lakewood, Colorado
  - Hope Hospice and Palliative Care, Fort Myers, Florida
  - LifePath Hospice and Palliative Care, Inc., Tampa, Florida
  - Hospice Care in the Berkshires, Inc., Pittsfield, Massachusetts
  - Hospice at Charlotte, Charlotte, North Carolina